CLINICAL TRIAL: NCT06639685
Title: Quantitative Mapping Based on Multi-parametric Functional MRI to Evaluate Renal Functions and Microstructure in Chronic Kidney Disease
Brief Title: Multi-parametric Functional MRI in Patients of Chronic Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-102
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease(CKD); MRI
Keywords: Chronic Kidney Disease; MR Fingerprinting; ASL
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD: Chronic Kidney Disease
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MR Fingerprinting and ASL

SUMMARY:
To explore the value of MR Fingerprinting-generated quantitative maps combined with ASL renal perfusion imaging in the assessment of renal impairment in chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) has become an important public health problem threatening human health worldwide. The prevalence rate of CKD in Chinese adults is 10.8%, but the awareness rate and diagnosis rate are generally low. At present, the assessment of renal impairment in CKD mainly relies on laboratory tests, such as estimated glomerular filtration rate (eGFR) and urinary protein/creatinine ratio, and the value of functional MRI in the assessment of renal impairment in patients with CKD is unclear. As a new sequence still in the scientific research stage, MR Fingerprinting can simultaneously generate quantitative T1 maps, T2 maps and proton-weighted images in one breath holding scan, with short scanning time, high repeatability and accuracy. It has been proved that quantitative techniques of T1 mapping and T2 mapping are valuable for evaluating the degree of renal fibrosis and water content. Kidney is a blood-rich organ, and the blood flow of kidney is of great significance to the evaluation of renal function. ASL uses hydrogen protons in arterial blood as an endogenous tracer to evaluate tissue blood perfusion, and can quantitatively evaluate renal blood perfusion in patients with CKD without the use of exogenous contrast agents, avoiding the risk of aggravated renal damage and nephrogenic fibrosis caused by injection of gadoline-containing contrast agents. The objective of our study was to explore the value of MRF sequence-generated quantitative maps combined with ASL renal perfusion imaging in the assessment of renal impairment in chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic kidney disease (CKD) by renal biopsy

Exclusion Criteria:

* Patients with serious underlying diseases
* Patients with MRI incompatible metal implants and contraindications such as claustrophobia
* Patients with imperfect clinical data and pathological data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with chronic kidney disease by renal biopsy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
T1 and T2 value | 3 months
  T1 and T2 value generated by MR Fingerprinting

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No